CLINICAL TRIAL: NCT02606032
Title: Randomized Trial of Antimicrobials Versus Placebo in Addition to Fecal Microbiota Therapy in for the Induction of Remission in Active Ulcerative Colitis
Brief Title: Trial of Antimicrobials Versus Placebo in Addition to Fecal Transplant Therapy in Ulcerative Colitis
Acronym: FMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Hamilton Academic Health Sciences Organization (Other)
Responsible Party: Principal Investigator, Paul Moayyedi, Director Division of Gastroenterology, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB# 0163
Record Dates: First submitted 2015-11-13; First posted 2015-11-17 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Ulcerative Colitis
Keywords: Fecal Microbiota Transplant; Antibiotics
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Metronidazole; Doxycycline; Terbinafine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metronidazole+doxycylcine+terbinafine (Active Comparator): Metronidazole 500 mg BID, Doxycycline 100 mg BID, Terbinafine 250 mg once daily all for 14 days
  Interventions: Drug: Metronidazole; Drug: Doxycycline; Drug: Terbinafine
- Placebo (Placebo Comparator): Placebo Metronidazole, Placebo Doxycycline, and Placebo Terbinafine all BID for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metronidazole — active comparator
  Other Names: Flagyl
  Arms: Metronidazole+doxycylcine+terbinafine
Drug: Doxycycline — active comparator
  Other Names: Vibramycin
  Arms: Metronidazole+doxycylcine+terbinafine
Drug: Terbinafine — active comparator
  Other Names: Lamisil
  Arms: Metronidazole+doxycylcine+terbinafine
Drug: Placebo — identical placebos to all antibiotics
  Arms: Placebo

SUMMARY:
The investigators will test the hypothesis that giving antibiotics prior to fecal transplant therapy for active UC increases the proportion of patients in remission at the end of treatment. The investigators will randomize patients aged 18 or over with active UC to antibiotics (metronidazole 500mg, doxycycline 100mg, Terbinafine 250 mg, all twice daily for two weeks); or identical placebo. At the end of two weeks the investigators will give all patients fecal transplant therapy twice per week for eight weeks from an anonymous donor stool.). Patients will complete a validated UC questionnaire, have a flexible sigmoidoscopy to assess the degree of inflammation in the colon and complete general and disease specific quality of life questionnaire as well as a questionnaire on anxiety and depression. Patients will complete the same questionnaires again at the end of treatment at week 9 when they will also have a repeat flexible sigmoidoscopy. The main outcome that will be assessed is the proportion of patients in remission from their UC at the end of treatment.

DETAILED DESCRIPTION:
Patients aged 18 or over with active UC defined as a Mayo score > 3 with an endoscopic score >0 will be eligible for the study. Subjects will be excluded if they are participating in another clinical trial, are unable to give informed consent, have severe comorbid medical illness, have concomitant Clostridium difficile infection or have severe UC requiring hospitalization. Continued treatment with 5-ASA, azathioprine, 6-mercaptopurine or anti-TNFα therapy (e.g. infliximab) will be permitted if taken at stable dose for ≥12 weeks prior to randomization. Eligible patients will be randomized 1:1 to metronidazole 500mg bid, doxycycline 100mg bid, Terbinafine 250 mg and or identical placebos all for two weeks. Patients will all then receive their first FMT 1-3 days after completing their course of antibiotic/placebo. FMT will be administered twice per week for 8 weeks.

Eighty active UC patients will be randomized 1:1 according to a computer generated randomization list. Randomization will be administered centrally at the GI Clinical Trials Unit to ensure concealment of allocation.

Subjects will have a sigmoidoscopy (or colonoscopy if clinically indicated), physician assessment and complete a Mayo score, IBDQ questionnaire, EQ5D and HAD questionnaires at baseline. A repeat sigmoidoscopy, Mayo score, IBDQ, EQ5D and HAD questionnaires will be completed at 9 weeks, at exit from the study (one week after last FMT). No new medical therapies (e.g. corticosteroids, antibiotics, probiotics) will be permitted during the 9 week study period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 or over
2. Active UC defined as a Mayo score > 3
3. A Mayo endoscopic score > 0

Exclusion Criteria:

1. Participating in another clinical trial
2. Unable to give informed consent
3. Severe co-morbid medical illness
4. Concomitant Clostridium difficile infection
5. Severe UC requiring hospitalization.
6. Increase in medical therapy for UC in the last 12 weeks. Continued treatment with 5-ASA, azathioprine, 6-mercaptopurine or anti-TNF alpha therapy (e.g. infliximab) will be permitted if taken at stable dose for ≥12 weeks prior to randomization. Relapse on a stable dose (same dose for at least 2 weeks) or a tapering dose of steroids will also be permitted provided the dose of steroid is not increased again. Stable intake of probiotic therapy also permitted.
7. Antibiotic therapy in the last 30 days.
8. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the randomized trial is remission of UC defined as a Mayo score < 3 with an endoscopic Mayo score = 0 at the end of the trial Transplant Therapy in Ulcerative Colitis | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Moayyedi, MD, Principal Investigator — Hamilton HSC
Locations (1):
- Hamilton Health Sciences / McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No